CLINICAL TRIAL: NCT04362696
Title: Improving Working Memory in Older Adults by Restoring Large-Scale Cortical Interactions
Brief Title: Improving Working Memory in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University Charles River Campus (Other)
Responsible Party: Principal Investigator, Robert Reinhart, Assistant Professor, Boston University Charles River Campus
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 4230E
Record Dates: First submitted 2020-04-21; First posted 2020-04-27 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Large-scale Physiological Foundations of Memory Decline in Aging Humans

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- active stimulation (Experimental)
  Interventions: Device: High definition transcranial electrical current stimulation
- sham stimulation (Sham Comparator)
  Interventions: Device: High definition transcranial electrical current stimulation

INTERVENTIONS:
Device: High definition transcranial electrical current stimulation — Low-intensity and safe, noninvasive application of electrical current to the human scalp with the goal of gradually modulating levels of neuronal excitability.

SUMMARY:
The research program will evaluate the theoretical claim that age-related memory and cognitive decline in humans result from the inefficient orchestration of rhythmic activity within large-scale cortical networks. The results will contribute to the basic science groundwork for developing future non-pharmacological interventions aimed at boosting memory and cognition in aging and clinical populations.

DETAILED DESCRIPTION:
We hypothesize that aged-related memory and cognitive impairments emerge from large-scale functional dysconnectivity, and by stimulating the brain noninvasively with extremely weak levels of electrical current, we may be able to re-synchronize connectivity and stabilize or improve memory and cognitive function, measured behaviorally. The experiments of this project are proposed as between-subjects, sham-controlled, and double-blind in design, and use noninvasive electroencephalographic (EEG) measurements of rhythmic brain activity. The experimental intervention involves the application of low-intensity, high-definition, transcranial electrical current stimulation while subjects perform a variety of computer-based tasks that probe memory and cognitive function.

ELIGIBILITY:
The following general inclusion criteria apply to all subjects: must be between the ages of 68-80 (except for Experiment 1 where subjects must be between the ages of 18-30), have normal or corrected-to-normal vision, color vision, nonpregnant, no metal implants in head, no implanted electronic devices, no history of neurological problems or head injury, no skin sensitivity, no claustrophobia, no dementia (normal Mini Mental State Examination between 24-30; Montreal Cognitive Assessment > 25), no depression (normal Beck Depression Inventory II <13; Geriatric Depression Scale < 10), and cannot be taking any psychoactive medication.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 964 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Memory performance success (sham stimulation condition) | During sham intervention
  The accuracy of task performance (in percentage correct units) in the delayed-match-to-sample working memory paradigm
Memory performance success (active stimulation condition) | During active intervention
  The accuracy of task performance (in percentage correct unit) in the delayed-match-to-sample working memory paradigm
Memory performance speed (sham stimulation condition) | During sham intervention
  The reaction time of task performance (in millisecond units) in the delayed-match-to-sample working memory paradigm
Memory performance speed (active stimulation condition) | During active intervention
  The reaction time of task performance (in millisecond units) in the delayed-match-to-sample working memory paradigm

CONTACTS AND LOCATIONS:
Locations (1):
- 677 Beacon St. Room 308, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No